CLINICAL TRIAL: NCT02578758
Title: The Differential Efficacy of a Specific Positive Psychology Components in a Transdiagnostic Internet-based Protocol for the Treatment of Emotional Disorders
Brief Title: Efficacy of a Transdiagnostic Internet-based Protocol in Community Sample
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UJAUMEI014
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Emotional Disorders; Anxiety; Depression
Keywords: Transdiagnostic Internet-based Protocol; Positive affect regulation
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Transdiagnostic Internet-Based Protocol (Experimental): Intervention group that carries out the Transdiagnostic Internet-Based Protocol and receives support by the therapist (a brief weekly two-minute phone call without clinical content and two weekly orientative text messages).
  Interventions: Behavioral: Transdiagnostic internet-based protocol
- Transdiagnostic Internet-Based Protocol+Positive Affect (Experimental): Intervention group that carries out the Transdiagnostic Internet-Based Protocol+Positive Affect component and receives support by the therapist (a brief weekly two-minute phone call without clinical content and two weekly orientative text messages).
  Interventions: Behavioral: Transdiagnostic internet-based protocol + positive affect component
- Waiting List Control Group (Other): Participants in a 18-week waiting list control condition. They will be offered the possibility of receiving the online treatment protocol after the waiting list period.
  Interventions: Other: Waiting List Control Group

INTERVENTIONS:
Behavioral: Transdiagnostic internet-based protocol — Transdiagnostic internet-based protocol is an Internet-based Protocol for ED, which will allow the individual to learn and practice adaptive ways to regulate their emotions from a transdiagnostic perspective. The protocol contains the following components: present-focused emotional awareness, cognitive flexibility, emotional avoidance and emotion-driven behaviors, interoceptive and situation-based emotion exposure, psychoeducation about emotions, motivational enhancement and relapse prevention, which are organized in 12 modules: Emotional disorders and emotion regulation; Motivation for change; Understanding the role of emotions; The acceptance of emotional experiences; Practicing the acceptance; Learning to be flexible; Practicing the cognitive flexibility; The emotional avoidance; Emotion driven behaviors; Accepting and facing physical sensations; Facing emotions in the contexts in which they occur; and Relapse Prevention.
  Arms: Transdiagnostic Internet-Based Protocol
Behavioral: Transdiagnostic internet-based protocol + positive affect component — Transdiagnostic internet-based protocol + positive affect component is an Internet-based protocol for ED. This protocol contains several transdiagnostic components (present-focused emotional awareness, cognitive flexibility, emotional avoidance and emotion-driven behaviors, interoceptive and situation-based emotion exposure, psychoeducation about emotions, motivational enhancement and relapse prevention) and a specific positive affect regulation component. These components are organized in 16 treatment modules: Emotional disorders and emotion regulation; Motivation for change; Understanding the role of emotions; The acceptance of emotional experiences; Practicing the acceptance; Learning to be flexible; Practicing the cognitive flexibility; The emotional avoidance; Emotion driven behaviors; Accepting and facing physical sensations; Facing emotions in the contexts in which they occur; Learning to move on; Learning to enjoy; Learning to live; Living and learning; and Relapse Prevention.
  Arms: Transdiagnostic Internet-Based Protocol+Positive Affect
Other: Waiting List Control Group — Participants in a 18-week waiting list control condition. They will be offered the possibility of receiving the online treatment protocol after the wating list period.
  Arms: Waiting List Control Group

SUMMARY:
The aim of this study is to assess the efficacy of a Transdiagnostic Internet-based Protocol (Emotion Regulation Protocol) for the treatment of Emotional Disorders (ED) (major depression disorder, dysthymic disorder, obsessive-compulsive disorder and four anxiety disorders: panic disorder, agoraphobia, generalized anxiety disorder, and social anxiety disorder) both in terms of efficacy regarding depressive and anxiety symptomatology and its potential impact on higher-order psychological dimensions (neuroticism/behavioral inhibition and low positive affect/behavioral activation) in a community sample. It will also be tested the differential effect of a specific treatment component based on positive psychology techniques in positive affect. The main hypotheses are: 1) both modalities of the protocol (TP and TP+PA) will be more effective than the WL condition in the primary outcome measures. Investigators also expect scores on positive affect to be higher in the TP+PA condition than in the TP condition.

DETAILED DESCRIPTION:
Emotional disorders (ED) (anxiety and mood disorders) are among the most prevalent mental disorders, with a life prevalence of 29% and comorbidity rates that range between 40 and 80%. If they are not adequately treated the course is often chronic, and significantly affect important functioning areas such as work and social relationships. Thus, these data strongly suggest efficacious and efficient treatments are needed in order to address this important health problem. The classification and differentiation of mental disorders carried out in manuals like the Diagnositc and Statistical Manual of Mental Disorders (DSM) and the International Classification of Diseases (ICD) has played an important role in the emphasis placed on the research about the treatment of specific disorders; however, it has also been a problem in the dissemination of evidenced-based treatments due to the difficulties in training the clinicians in the variety of the available disorder-specific programs. In the other hand, Evidence-based psychological treatments (EBPT) have shown efficacy in the treatment of ED, however, less than 50 % of people with ED receive treatment and causes include costs, time of application and the lack of well-trained professionals. In addition, epidemiological studies have shown that at least 55% of people suffering from an anxiety disorder suffer from another anxiety disorder at the moment of the assessment, and this prevalence rate is up to 76% when different lifespan diagnoses are taken into account. This high comorbidity rate indicates that the different ED share important characteristics and it has been proposed that this overlapping is accounted for by common biological and psychological vulnerabilities that along with psychosocial stress factors leads to different manifestations of the same vulnerability, i. e., the different mood and anxiety disorders. Thus, a Transdiagnostic approach could help overcome these barriers.

Transdiagnostic approaches have implications in the treatment of psychological disorders as a number of treatment protocols have been developed based on this perspective. Clark has distinguished three perspectives in transdiagnostic cognitive-behavioral therapy: a) The transdiagnostic practice, a pragmatic perspective that includes components of various disorder-specific intervention protocols whose aim is to determine which are the active components in samples with those disorders. The contributions of Norton, Andrews and Titov, and the study: Coordinated Anxiety Learning and Management (CALM) belong to this category. b) The transdiagnostic theory, that specifies a theoretical framework which outlines the common psychological constructs that influence the maintenance of ED. For instance, the tripartite model of anxiety and depression, with positive and negative affect as relevant constructs. c) The Unified Protocol. The Barlow's team has designed a protocol, adequate for the treatment of ED which focuses on four essential aspects: to increase present-focused emotional awareness, to identify and modify emotional avoidance patterns, to promote the cognitive flexibility and to facilitate exposure to avoided situations and sensations.

Another aspect that could enhance the dissemination of evidence-based treatments as well as considerably reduce the costs is the use of the Internet. A number of systematic reviews has shown that Internet-based treatments yield similar results when compared to face-to-face therapy. Nevertheless, most of these programs are focused on a single disorder since very few transdiagostic internet-based treatments have been developed and tested by means of randomized controlled trials so far.

The main objective of the treatment components of the Unified Protocol (UP) is to train patients in the regulation of negative emotions or negative affect (NA), but less attention has been paid to the inclusion of treatment components directly targeting positive affect (PA) regulation.

Investigators of this research group (LabPsiTec) have developed a traditional transdiagnostic treatment that is partly based on the UP and it has been added a specific component of positive affect regulation in order to more directly target the regulation of positive affect. The study will include three conditions: 1) Transdiagnostic protocol (TP); 2) Transdiagnostic protocol + positive affect component (TP+PA); and 3) Waiting list control group (WL).

The main hypothesis is that both modalities of the protocol (TP and TP+PA) will result more effective than the WL condition in the primary outcome measures. Investigators expect scores on positive affect to be higher in the TP+PA condition than in the TP condition.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years old or older.
* Meeting the DSM-IV diagnosis criteria of emotional disorder (panic disorder, agoraphobia, social anxiety disorder, generalized anxiety disorder, obsessive-compulsive disorder, major depression disorder and dysthymia).
* Providing written, informed consent.
* Being able to understand and read Spanish.
* Having daily access to the Internet in their natural environment.

Exclusion Criteria:

* Being diagnosed a severe mental disorder (people with the following mental disorders will be excluded from the study: schizophrenia, bipolar disorder and personality disorders from clusters A and B).
* Being diagnosed an alcohol and/or substance dependence disorder.
* The presence of high suicidal risk.
* A medical disease or condition which prevent the participant from carry out the psychological treatment.
* Receiving another psychological treatment while the study is still ongoing.
* The increase and/or changes in the medication of participants receiving pharmacological treatment during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2014-09; Primary Completion 2019-11 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in the Beck Depression Inventory II (BDI-II) (Beck, Steer, & Brown, 1996) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  The BDI-II is one of the most widely used questionnaires to evaluate the severity of depression in pharmacological and psychotherapy trials. It consists of 21 items about the different symptoms characterizing the major depression disorder, summed to obtain the total score, which can be a maximum of 63 points. The instrument has good internal consistency (Cronbach's alpha of 0.76 to 0.95) and a test-retest reliability of around 0.8.
Change in the Beck Anxiety Inventory (BAI) (Beck, & Steer, 1990) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  The BAI is a 21-item self-report measure designed to assess anxiety. Each item has a 4-point Severity scale (e.g., not at all, mildly, moderately, and severely) that addresses symptoms experienced during the past week. The internal consistency of the BAI has been found to range from .85 to .94 and has been found to have adequate convergent and divergent validity.

SECONDARY OUTCOMES:
Change in the Obsessive-Compulsive Inventory (OCI-R) (Foa et al., 2002) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  The OCI-R is a scale made up of 18 items rated 1 to 4 and organized in 6 dimensions (washing, verification, order, obsession, hoarding and mental neutralization) that assesses obsessive-compulsive behaviors. The OCI-R has a good internal consistency (coefficient alpha between .81 and .93), a good to excellent test-retest reliability (between .57 and .91), a good convergent validity and a solid factor structure.
Change in the Self-Reported Panic Disorder Severity Scale (PDSS-SR) (Houck, Spiegel, Shear, & Rucci, 2002) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  The scale measures the severity of the panic disorder through measures of panic attack frequency, distress during the panic attacks, anticipatory anxiety, fear and agoraphobic avoidance, fear and avoidance of physical sensations, and work and social impairment. The reliability of the scale has proved to be excellent (coefficient alpha of .917) as also has done the test-retest reliability (ICC = .81).
Change in the Pen State Worry Questionnaire (PSWQ) (Meyer, Miller, Metzger, & Borkovec, 1990) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  It is a questionnaire that evaluates the worry as an incontrollable, generalized and excessive experience. The psychometric properties of the PSWQ have proved to be good, with an internal consistency ranging from .91 to .95, and a good validity and test-retest reliability.
Change in the Social Interaction Anxiety Inventory (SIAS) (Mattick y Clarke, 1998) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  This scale is made up of twenty items rated 0 to 4 that asses the anxiety experienced by the patient in social interactive situations. The scale has a good internal consistency (alpha coefficient between .88 and .94), good test-retest and discriminant reliability, as well as appropriate construct validity.
The Positive and Negative Affect Schedule (PANAS) (Watson, Clark y Tellengen, 1988; Sandín et al., 1999) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  The PANAS consists of 20 items that evaluate two independent dimensions: positive affect (PA) and negative affect (NA). The range for each scale (10 items on each) is from 10 to 50. The Spanish version has demonstrated high internal consistency (α = 0.89 and 0.91 for PA and NA in women, respectively, and α = 0.87 and 0.89 for PA and NA in men, respectively) in college students.

OTHER OUTCOMES:
Quality of Life Index (QLI) (Mezzich et al., 2000) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  It consists of 10 items that evaluate perceived well-being in different areas (physical, psychological/emotional, occupational functioning, interpersonal functioning, among others). The test-retest reliability correlation coefficient of the Spanish version of the QLI mean score was .89.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Botella, Professor, Study Director — Universitat Jaume I, Castellon, Spain; Amanda Díaz, PhD Student, Study Chair — Universitat Jaume I, Castellon, Spain
Locations (1):
- Universitat Jaume I, Castellon, Castelló, Spain

REFERENCES:
- [Background] Titov N, Andrews G, Johnston L, Robinson E, Spence J. Transdiagnostic Internet treatment for anxiety disorders: A randomized controlled trial. Behav Res Ther. 2010 Sep;48(9):890-9. doi: 10.1016/j.brat.2010.05.014. Epub 2010 May 24. PMID 20561606
- [Background] Titov N, Dear BF, Schwencke G, Andrews G, Johnston L, Craske MG, McEvoy P. Transdiagnostic internet treatment for anxiety and depression: a randomised controlled trial. Behav Res Ther. 2011 Aug;49(8):441-52. doi: 10.1016/j.brat.2011.03.007. Epub 2011 Apr 3. PMID 21679925
- [Background] Farchione TJ, Fairholme CP, Ellard KK, Boisseau CL, Thompson-Hollands J, Carl JR, Gallagher MW, Barlow DH. Unified protocol for transdiagnostic treatment of emotional disorders: a randomized controlled trial. Behav Ther. 2012 Sep;43(3):666-78. doi: 10.1016/j.beth.2012.01.001. Epub 2012 Jan 18. PMID 22697453
- [Background] Carl JR, Soskin DP, Kerns C, Barlow DH. Positive emotion regulation in emotional disorders: a theoretical review. Clin Psychol Rev. 2013 Apr;33(3):343-60. doi: 10.1016/j.cpr.2013.01.003. Epub 2013 Jan 12. PMID 23399829
- [Derived] Diaz-Garcia A, Gonzalez-Robles A, Garcia-Palacios A, Fernandez-Alvarez J, Castilla D, Breton JM, Banos RM, Quero S, Botella C. Negative and Positive Affect Regulation in a Transdiagnostic Internet-Based Protocol for Emotional Disorders: Randomized Controlled Trial. J Med Internet Res. 2021 Feb 1;23(2):e21335. doi: 10.2196/21335. PMID 33522977
- [Derived] Diaz-Garcia A, Gonzalez-Robles A, Fernandez-Alvarez J, Garcia-Palacios A, Banos RM, Botella C. Efficacy of a Transdiagnostic internet-based treatment for emotional disorders with a specific component to address positive affect: Study protocol for a randomized controlled trial. BMC Psychiatry. 2017 Apr 20;17(1):145. doi: 10.1186/s12888-017-1297-z. PMID 28424068
- See also: Laboratory of Psychology and Technology of the University Jaume I — http://www.labpsitec.uji.es
- See also: Web site of the intervention program — http://www.psicologiaytecnologia.com